CLINICAL TRIAL: NCT05819580
Title: Mesothelioma Clinical Trials Review: Examining Patient Experiences in Mesothelioma Clinical Trials to Identify Influencing Factors
Brief Title: Studying the Clinical Trial Experiences of Patients With Mesothelioma
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80693772
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Mesothelioma
Keywords: mesothelioma
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medical research participation percentages haven't always been fully representative of a given demographic.

The goal is to find out which aspects of a clinical study may make it more difficult for patients to take part or see it through.

The data will be evaluated through different demographic lenses and identify trends that could help improve the experience of future mesothelioma patients during clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Must have a medical diagnosis of mesothelioma that has been confirmed by a physician.
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Pregnant or lactating woman
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mesothelioma patients who are actively considering involvement in an observational clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a mesothelioma medical study. | 3 months
Number of mesothelioma patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sinn K, Mosleh B, Hoda MA. Malignant pleural mesothelioma: recent developments. Curr Opin Oncol. 2021 Jan;33(1):80-86. doi: 10.1097/CCO.0000000000000697. PMID 33186182
- [Background] Jakobsen JN, Sorensen JB. Review on clinical trials of targeted treatments in malignant mesothelioma. Cancer Chemother Pharmacol. 2011 Jul;68(1):1-15. doi: 10.1007/s00280-011-1655-3. Epub 2011 May 7. PMID 21553148
- [Background] Lau B, Boyer M, Lee JH, Kao S. Clinical Trials Eligibility of Patients With Malignant Pleural Mesothelioma: Use of Novel Therapies and Outcomes. Clin Lung Cancer. 2020 Jul;21(4):378-383.e1. doi: 10.1016/j.cllc.2020.01.007. Epub 2020 Mar 7. PMID 32249197

DOCUMENTS (1):
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT05819580/ICF_000.pdf